CLINICAL TRIAL: NCT06492642
Title: Pilot Study of Personalized Patient Education for Chronic Low Back Pain
Brief Title: Research Study on Patient Education for People With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Allyn Bove, Assistant Professor of Physical Therapy, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24020023
Record Dates: First submitted 2024-06-21; First posted 2024-07-09 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic Low-Back Pain; Patient Education
MeSH Terms: interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: 20 individuals with chronic low back pain. Will aim to recruit a socioeconomically diverse sample. No randomization or group assignment; analyses will be conducted using a pre-post design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Education for Chronic Low Back Pain (Experimental): Patients will access online patient education materials on chronic low back pain five times after completing baseline questionnaires on days 5, 8, 11, 14, and 17.
  Interventions: Other: Patient Education for Chronic Low Back Pain

INTERVENTIONS:
Other: Patient Education for Chronic Low Back Pain — Patient education on chronic low back pain (LBP), including:
  Day 5: Basic LBP education, types of LBP, "red flags"; Day 8: LBP guideline recommendations re: imaging; Day 11: LBP guideline recommendations re: use of rehabilitation services, sitting and standing desks; Day 14: LBP guideline recommendations re:pharmacologic management; Day 17: LBP guideline recommendations re: injections and surgery.

SUMMARY:
The goal of this pilot single-arm study is to examine the potential of personalized patient education materials to improve self-efficacy and perceived functional disability in patients with chronic low back pain. The main questions it aims to answer are:

1. What is the feasibility of delivering a personalized patient education program for individuals with chronic low back pain?
2. What is the impact of personalized patient education materials on disease-specific self-efficacy and patient-reported function in a small sample of individuals with chronic low back pain?

Participants will be asked to:

* access and complete online baseline questionnaires
* access and follow online patient materials on chronic low back pain on days 5, 8, 11, 14, and 17
* access and complete online follow-up responses to baseline questionnaires and a post-study survey

DETAILED DESCRIPTION:
This is a pilot single-arm study to examine the potential of personalized patient education materials to improve self-efficacy and perceived functional disability for patients with chronic low back pain (cLBP).

The investigators aim to recruit 30 individuals with cLBP. The investigators will aim to recruit 15 individuals from areas with an Area Deprivation Index (ADI) of at least 6 and 15 from areas with an ADI of 5 or lower.

Participants will complete a 3-week educational intervention aimed at improving self-efficacy in managing chronic LBP. Educational materials will be personalized for each participant depending upon things like baseline knowledge of cLBP, smoking status, exercise status, beliefs about safe movement with cLBP, preference for various health care interventions, and nature of work (sedentary vs. labor-oriented job).

Educational materials will be provided electronically using Qualtrics.

Participants will complete outcome measures at baseline and follow-up as described elsewhere in this study record.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Existence of chronic low back pain, defined as back pain that has lasted longer than 12 weeks
* Has sought care for LBP within the past 12 months, confirmable through medical records
* Classified as having at least "moderate" LBP-related disability, defined as a raw score of 15 or higher (out of 50) on the Oswestry Disability Index (additional detail below in Outcomes) upon telephone screening

  * Patients who receive care through UPMC: The study team will confirm in Epic that the participant has indeed had a health care encounter that included a diagnosis of low back pain in the previous 12 months
  * Patients who receive care outside of UPMC: The potential participant can provide a physician letter, after visit summary, or other reasonable documentation to confirm that they have indeed sought health care for LBP within the previous 12 months
* (for 50% of participants) Area Deprivation Index (ADI) of 6 or higher, using the Pennsylvania-specific deciles. The investigators will use ADI as a marker of socioeconomic status. Although the sample size in this study will not be large enough to detect the ability of the intervention to reduce socioeconomic disparities in chronic LBP outcomes, the investigators do need to show that the investigators are able to recruit a sufficient population of individuals of lower socioeconomic status and individuals of higher socioeconomic status to demonstrate feasibility for a future larger study. State-level ADI is measured from 1 to 10, with lower scores indicating greater advantage, and higher scores indicating greater deprivation. It is measured at the level of a census block group. The investigators will identify a potential participant's ADI by inputting their address of residence into the Neighborhood Atlas mapping tool, which is freely available online at https://www.neighborhoodatlas.medicine.wisc.edu/mapping

Exclusion Criteria:

* any prior spine surgery
* any orthopaedic surgery in the past 6 months
* does not have own smartphone, tablet, laptop, or desktop to access study questionnaires and education materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Personal Pain Beliefs on Pain Self-Efficacy Questionnaire (PSEQ) at Day 21 | Baseline Day 0 & Day 21
  The PSEQ is a 10-item questionnaire that assesses an individual's confidence in performing specific functional activities despite ongoing pain. Reliability, validity, and internal consistency of the PSEQ have been established when used with patients with spine conditions. Possible scores range from 0-60 with higher scores indicating greater self-efficacy for managing pain.
  Change= (Day 21 score - Baseline score)
Feasibility of delivering a personalized patient education program for individuals with chronic low back pain - Recruitment | Through overall study completion, about 7 months
  - recruitment of at least 30 participants in 3 months
Feasibility of delivering a personalized patient education program for individuals with chronic low back pain - Retention | Through overall study completion, about 7 months
  - retention of at least 80% of those participants through follow-up data collection
Feasibility of delivering a personalized patient education program for individuals with chronic low back pain - Missing Data | Through overall study completion, about 7 months
  - missing data of no greater than 20% for any given data element

SECONDARY OUTCOMES:
Change from Baseline Subjective Level of Disability on Oswestry Disability Index (ODI) at Day 21 | Baseline Day 0 & Day 21
  In addition to using the ODI as an eligibility screening tool, the investigators will also use it as a secondary outcome to measure patient-reported physical function relative to LBP. The ODI is a 10-item questionnaire that is considered the gold standard of LBP functional outcome assessments. Possible scores range from 0 to 100 with higher scores indicating more severe disability caused by LBP.
  Change= (Day 21 score - Baseline score)
Change from Baseline Pain on Numeric Pain Rating Scale (NPRS) at Day 21 | Baseline Day 0 & Day 21
  The NPRS is a one item, 11-point tool that simply asks the user to rate their pain on a whole-number scale from 0 to 10. The investigators will ask participants to rate their average LBP over the last 24 hours. Possible scores range from 0 (no pain at all) to 10 (worst imaginable pain).
  Change= (Day 21 score - Baseline score)

CONTACTS AND LOCATIONS:
Overall Officials: Allyn Bove, PhD, PT, DPT, Principal Investigator — University of Pittsburgh; Yanshan Wang, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share IPD with other researchers.

REFERENCES:
- [Background] Lewis M, Bromley K, Sutton CJ, McCray G, Myers HL, Lancaster GA. Determining sample size for progression criteria for pragmatic pilot RCTs: the hypothesis test strikes back! Pilot Feasibility Stud. 2021 Feb 3;7(1):40. doi: 10.1186/s40814-021-00770-x. PMID 33536076
- See also: Neighborhood Atlas Mapping Tool — https://www.neighborhoodatlas.medicine.wisc.edu/mapping

DOCUMENTS (1):
  • Informed Consent Form (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT06492642/ICF_000.pdf